CLINICAL TRIAL: NCT06867562
Title: A Phase-3, Randomized, Parallel Group, Open-label, Multicenter, Two-Arm Treatment Study to Evaluate the Efficacy and Safety of Weekly Paclitaxel Lipid Suspension Compared with Weekly Conventional Paclitaxel in the Patients with Platinum-Resistant/Refractory Recurrent High-grade Serous Epithelial Ovarian Cancer Including Fallopian Tube And/or Primary Peritoneal Cancer
Brief Title: Paclitaxel Lipid Suspension for Patients with Platinum-Resistant /Refractory Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jina Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0127-23
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Platinum-Resistant Primary Peritoneal Carcinoma; Platinum Resistant High Grade Epithelial Ovarian Cancer; Platinum Resistant High Grade Serous Ovarian Cancer
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Intervention Model Description: At baseline, participants will be randomized to either the Paclitaxel Lipid Suspension arm or the Conventional Paclitaxel arm. Participants in both arms will continue the treatment till either disease progression as assessed by investigator. Disease status and tumor response will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST v1.1) and Gynecologic Cancer Intergroup (GCIG) Cancer Antigen 125 guidelines. To ensure consistent interpretation of measurable disease and objective endpoints for the study, all imaging studies performed throughout the study will be sent to a blinded independent central review (BICR) vendor for tumor measurement and evaluation of response.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paclitaxel Lipid Suspension for Injection (Experimental): Participants will be administered Paclitaxel Lipid Suspension infusion at a dose of 80 mg/m2 for over 1 hour on days 1, 8 and 15 of each cycle. The cycle length for the Paclitaxel Lipid Suspension weekly schedule is 28 days.
  Interventions: Drug: Paclitaxel Lipid Suspension
- Conventional paclitaxel (Active Comparator): Participants will be administered Conventional Paclitaxel infusion at a dose of 80 mg/m2 for over 1 hour on days 1, 8 and 15 of each cycle. The cycle length for the Paclitaxel Lipid Suspension weekly schedule is 28 days.
  Interventions: Drug: Conventional paclitaxel or Taxol

INTERVENTIONS:
Drug: Paclitaxel Lipid Suspension — The formulation consists of uniformly sized (< 100 nm) particles of Paclitaxel suspended in a lipid-based formulation. The advantage of such a Lipid-Based formulation of Paclitaxel is an improvement of the safety profile by eliminating excipients, Cremophor and ethanol which are present in conventional Paclitaxel formulations (Taxol®).
  Arms: Paclitaxel Lipid Suspension for Injection
Drug: Conventional paclitaxel or Taxol — Conventional formulation with detergent Cremophor and alcohol
  Arms: Conventional paclitaxel

SUMMARY:
This is a phase-3, open-label, multicenter, two-arm treatment study to evaluate the efficacy and safety of weekly Paclitaxel Lipid Suspension compared with weekly conventional paclitaxel in participants with platinum-resistant/refractory recurrent high-grade serous epithelial ovarian cancer.

Paclitaxel Lipid Suspension or conventional paclitaxel will be administered intravenously at a dose level of 80 mg/m2 on Day 1, Day 8 and Day 15 of each 28 days cycle.

The primary objective is to establish the non-inferiority of Paclitaxel Lipid Suspension in comparison with conventional paclitaxel for Injection in participants with platinum-resistant/refractory recurrent advanced high-grade serous epithelial ovarian cancer including fallopian tube and/or primary peritoneal cancer.

Participants in both arms will be dosed with the drug until disease progression as assessed by investigator and/or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is willing to give written signed and dated informed consent to participate in the study.
2. Female ≥18 years of age fulfilling all other eligibility criteria.
3. Participants must have histopathologically/cytologically confirmed diagnosis of high-grade serous epithelial carcinoma of the ovary, fallopian tube cancer or primary peritoneal carcinoma. Non-epithelial or mixed (<50% of the primary tumor confirmed to be high-grade serous) epithelial/non-epithelial tumors (including malignant mixed Müllerian tumors), ovarian tumors with low malignant potential (borderline tumors), endometrioid, clear cell, mucinous or low-grade serous carcinomas or not otherwise specified (NOS) ovarian tumors are excluded.
4. Platinum resistant or refractory disease as per standard clinical and Gynecologic Oncology Group definition. Platinum-resistant/refractory disease is defined as disease progression within 6 months (182 days) following the last administered dose of platinum therapy (resistant), or lack of response or disease progression while receiving the most recent platinum-based therapy (refractory), respectively for whom single-agent paclitaxel is considered an acceptable therapeutic option by the investigator.
5. Participants must have received at least one-prior platinum-based chemotherapy regimen, including cisplatin, carboplatin or other organoplatinum compounds, for treatment of primary or recurrent ovarian, fallopian tube or primary peritoneal cancer.
6. Have at least one measurable lesion as per the RECIST criteria (version 1.1).
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
8. Left Ventricular Ejection fraction (LVEF) ≥50% as per Echocardiography (ECHO).
9. Participant has recovered from adverse events (baseline or ≤ CTCAE Grade 1) due to prior anti-cancer therapy(ies) (including surgery, radiotherapy, chemotherapy, targeted therapy, hormonal therapy) unless AE(s) is either clinically nonsignificant or stable on supportive therapy or do not constitute a safety risk to the participant as determined by the investigator.
10. Participants with life expectancy of at least 6 months in the Investigator's opinion.
11. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

    * Is not a woman of childbearing potential (WOCBP) OR
    * Is a WOCBP and agrees to remain on an acceptable contraceptive method that is highly effective (with a failure rate of <1% per year) for at least 6 months after the last dose of IMP.
    * A WOCBP agrees not to donate eggs (ova, oocytes) or freeze them for future use for reproduction during the recommended period of contraception. A WOCBP agrees to seek advice about the donation and cryopreservation of germ cells.
    * A WOCBP must have a negative highly sensitive serum pregnancy test at screening and a negative urine pregnancy test within 24 hours before the first dose of IMP.
    * If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required.
12. Participants with adequate bone marrow, renal and hepatic function
13. Has had prior PARP inhibitors for participants with documented breast cancer gene (BRCA) mutation (germline and/or somatic) or HRD status, unless the participant is not eligible for treatment with a PARP inhibitor due to precautions/intolerance, or if the treatment is not approved locally or not available due to any reasons.
14. Has had prior treatment with mirvetuximab soravtansine for participants with documented high folate receptor alpha expression, unless the participant is not eligible for treatment with mirvetuximab soravtansine due to precautions/intolerance, or if the treatment is not approved or available locally.
15. Participants must have progressed radiologically on or after their most recent line of systemic therapy. Biochemical progression will not be considered progression for this study.

Exclusion Criteria:

1. Have previously received paclitaxel at any time in the platinum-resistant setting. This does not apply to the participants who have received paclitaxel either in a neo/adjuvant setting in the first line or platinum-sensitive relapse.
2. Participants who are candidates for debulking surgery, or in whom chemotherapy is planned to shrink the otherwise inoperable tumor and make it operable even if the intent is palliative.
3. Participants who are planned to receive concurrent PARP inhibitors based on BRCA positivity and HRD status in line with approved indications of respective PARP inhibitors.
4. Participants who are using known strong CYP3A4 inducers, CYP3A4 inhibitors, CYP2C8 strong inhibitors, and strong inducers.
5. Participants who are planned for concurrent bevacizumab along with IMP for their disease management during the study. Participants who have received bevacizumab in the past for the management of ovarian cancer are eligible.

   Maintenance therapy (e.g., bevacizumab, PARP inhibitors) will be considered as part of the preceding line of therapy (i.e., not counted independently).
6. Participants with clinically significant current or recent (within the past 6 months before randomization) cardiac conditions as defined below:

   * Unstable angina
   * Myocardial infarction
   * Severe uncontrolled ventricular arrhythmias
   * Clinically significant pericardial disease
   * Electrocardiographic evidence of acute ischemia
   * Participants with evidence of abnormal cardiac conduction (e.g., bundle branch block or heart block) except in whom the disease has been stable
   * History of cardiac disease that met the NYHA Classification class 2 or greater
   * Cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism
7. Uncontrolled diabetes (defined as HbA1c ≥8% as per ADA) or has an active infection requiring systemic therapy.
8. History of drug or alcohol abuse according to medical history assessment by the investigator within 1 year before Screening or positive test result(s) for alcohol or drugs of abuse (including barbiturates, opiates, cocaine, cannabinoids, amphetamines and benzodiazepines) at Screening.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks before the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 28 days before trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
10. The receipt of an investigational medicinal product or participation in other drug research study within a period of 30 days before the first dose of an investigational medicinal product for the current study.
11. Pre-existing motor or sensory neurotoxicity of a severity ≥ grade 2 as defined by NCI CTCAE v5.0 criteria.
12. History of clinically significant liver or renal insufficiency; vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances that, in the investigator's judgment, might increase the risk to the participant or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study.
13. Participants who are unwilling or unable to follow protocol requirements.
14. Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years; carcinoma in situ of the cervix; or malignancy, which is considered cured with minimal risk of recurrence.
15. Prior known hypersensitivity reactions to and/or any of their excipients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 166 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate | Minimum 6 months
  The proportion of participants whose Best Overall Response is a confirmed CR or PR as determined by blinded independent central review (BICR) based on RECIST v1.1